CLINICAL TRIAL: NCT06504147
Title: A Phase 2, Randomised, Open Label, Multicentre Study of an Intraperitoneal α-emitting Radionuclide Therapy (Radspherin®) in Patients With Primary Advanced High-grade Serous or High-grade Endometrioid Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer, With Peritoneal Metastasis That Are Homologous Recombination Proficient and Scheduled to Undergo Neoadjuvant Chemotherapy and Interval Debulking Surgery
Brief Title: A Study of Radspherin® in Patients With Primary Advanced Epithelial Cancer, With Peritoneal Metastasis That Are Homologous Recombination Proficient Scheduled to Undergo Neoadjuvant Chemotherapy and Interval Debulking Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oncoinvent AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RAD-18-003
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Peritoneal Carcinomatosis; Ovarian Cancer
MeSH Terms: conditions — Peritoneal Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Radspherin (Experimental)
  Interventions: Drug: Radspherin
- Control (No Intervention)

INTERVENTIONS:
Drug: Radspherin — Radspherin® suspension consists of bio-degradable calcium carbonate micro particles with the α-emitting radionuclide 224Ra in suspension. 224Ra has a physical half-life of 3.6 days.
  Arms: Radspherin

SUMMARY:
This is a Phase 2, controlled, randomised, parallel assignment, open label, multicentre study to evaluate efficacy and safety of a single intraperitoneal injection of Radspherin® in patients with primary advanced high-grade serous or high-grade endometrioid epithelial ovarian cancer, fallopian tube, or primary peritoneal cancer, with peritoneal metastasis that are HR proficient and scheduled to undergo NACT and IDS. The study will be conducted in 2 parts; first, a Safety Lead-in Cohort will be recruited followed by the randomised part of the study. For both parts of the study, patients must be scheduled to undergo NACT and IDS and complete resection to no residual tumour (R0) should be deemed to be achievable during diagnostic work-up. Patients in both parts of the study will undergo the same procedures and assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent and to comply with the clinical study protocol (CSP).
2. Female of age ≥ 18 years.
3. Patients with primary advanced high-grade serous or high-grade endometrioid epithelial ovarian, fallopian tube, or primary peritoneal cancer (FIGO Stage IIIB/C or IV).
4. Peritoneal and other metastases eligible for IDS to no residual tumour.
5. Adverse events recovered to at least Grade 1 from the effects (excluding alopecia) of any prior medical therapy for malignancy.
6. Confirmed HR proficient by Myriad MyChoice CDx testing.
7. Received NACT (numbers of cycles as per investigator's discretion) with regress or stable disease on diagnostic imaging and assessed to be operable to R0 pre-surgery.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status Score of 0 to 2 and patient fit enough to undergo IDS and further treatment according to standard of care.
9. Adequate renal function:

   • Calculated creatinine clearance using the Cockcroft-Gault formula ≥ 40 ml/min or measured creatinine clearance ≥ 40 ml/min.
10. Adequate hepatic function:

    * Serum bilirubin < 1.5 x upper limit of normal (ULN), and
    * Aspartate transaminase and alanine transaminase ≤ 3 x ULN.
11. Adequate bone marrow function:

    * Absolute neutrophil count ≥ 1.0 x 10^9/l, and
    * Platelets ≥ 100 x 10^9/l, and
    * Haemoglobin ≥ 9 g/dL.
12. For females of childbearing potential, a negative pregnancy test must be documented prior to enrolment.
13. For females of childbearing potential agreement to use at least one of the following highly effective (failure rate < 1%) methods of contraception during the treatment period and for at least 9 months if they receive Radspherin®, unless hysterectomy or oophorectomy is performed during IDS.

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient), periodic abstinence (e.g. calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Female sterilisation (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least 6 weeks before enrolment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    * Use of oral (oestrogen and progesterone), injected or implanted hormonal methods of contraception or placement of an intrauterine device or intrauterine system, or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception. In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

Note: In addition to the use of one highly effective method of contraception as listed above, a condom is required for all male partners during the treatment period and for at least 9 months after the dose of IMP, unless vasectomised at least 6 months prior to enrolment.

Exclusion Criteria:

1. Known somatic or germline BRCA1 or BRCA2 mutations or confirmed HR deficient.
2. Suspicion of peritoneal leak, shunt, or otherwise suspected atypical target compartment pharmacokinetics, based on investigator's judgement, patient history and diagnostic images.
3. Epithelial borderline tumours, ovarian clear cell carcinoma, mucinous ovarian carcinoma, malignant Brenner tumours, non-epithelial ovarian malignancies, carcinosarcoma and neuroendocrine tumours or recurrent ovarian cancer.
4. Symptomatic central nervous system metastasis.
5. Another primary malignancy within the past 3 years (except for non melanoma skin cancer, cutaneous melanoma stage 1, cervical cancer in situ or FIGO 2023 Stage IA1 or IA3 prior or synchronous endometrial cancer).
6. Prior abdominal/pelvic radiotherapy.
7. Disease progression during NACT.
8. Pregnant or lactating (nursing) women.
9. Active infections requiring antibiotics, and/or physician monitoring, or recurrent fever > 38.0⁰C associated with a clinical diagnosis of active infection.
10. Active liver disease with positive serology for active hepatitis B, hepatitis C or known human immunodeficiency virus (HIV).
11. Concurrent congestive heart failure or prior history of New York Heart Association (NYHA) class III/IV cardiac disease.
12. Any condition or illness that, in the opinion of the investigator or the medical monitor, would compromise the safety of the patients or interfere with the evaluation of the safety of the investigational medicinal product.
13. In the investigator's opinion not able to comply with study procedures. Any medical or psychological condition that would preclude participation in the study or compromise the ability to give informed consent.
14. Administration of an investigational medicinal product within 4 weeks, or at least 5 times the half life, prior to enrolment.
15. Concurrent administration of any cancer therapy other than planned study treatment within 4 weeks prior to, and up to 4 weeks after the surgery.
16. Treatment with bevacizumab within 5 weeks prior to IDS.
17. Known hypersensitivity to any of the excipients of the study drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 24 months
  To compare PFS in patients with primary advanced high-grade serous or high-grade endometrioid epithelial ovarian, fallopian tube, or primary peritoneal cancer1 with peritoneal metastasis that are HR proficient following Radspherin® treatment versus no treatment.

SECONDARY OUTCOMES:
Peritoneal progression free survival | 24 months
  To compare peritoneal PFS (PPFS) in patients with primary advanced epithelial cancer with peritoneal metastasis that are HR proficient following Radspherin® treatment versus no treatment.

CONTACTS AND LOCATIONS:
Locations (10):
- Moffitt Cancer Center, Tampa, Florida, United States
- UZ Leuven, Leuven, Belgium
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy
- The Norwegian Radiumhospital, Oslo, Norway
- Spain (4):
  - Hospital Universitari de Bellvitge, Barcelona
  - Clinica Universidad de Navarra, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitari i Politècnic La Fe, Valencia
- United Kingdom (2):
  - Imperial College Healthcare NHS Trust, London
  - University Hospital Southampton NHS Foundation Trust, Southampton